CLINICAL TRIAL: NCT06808256
Title: The Effect of Acupuncture on Hemodynamics and Pain of Post Craniotomy Patients With Mechanical Ventilation in the ICU of Tangerang Regency Hospital Banten
Brief Title: Effect of Acupuncture on Hemodynamics and Pain of Post Craniotomy Patients With Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Zellah Fransisca Natalia, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 24-12-1830
Record Dates: First submitted 2025-02-03; First posted 2025-02-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Post Craniotomy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The acupuncture therapy combined with standard therapy will be designated as the intervention group, while the standard therapy only will be designated as the control group
Who Masked: Outcomes Assessor
Masking Description: the outcome assessors will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The acupuncture and standard therapy
  Interventions: Procedure: the acupuncture therapy; Other: Standard therapy
- Control Group (Active Comparator): Standard therapy only
  Interventions: Other: Standard therapy

INTERVENTIONS:
Procedure: the acupuncture therapy — Acupuncture is performed for 3 consecutive days, using filiform needles in the chest, hands, feet area with 20 minutes retention during therapy and using press needle on the forehead which are retained for 3 days and after 3 days the stick needles will be removed. And patient continue to receive standard therapy in accordance with the clinical practice guidelines of the ICU Tangerang Hospital
  Arms: Intervention Group
Other: Standard therapy — Pharmacological therapy provided by the doctor in charge of anesthesia science patients to the research subjects was in accordance with existing clinical practice guidelines. In the ICU of Tangerang Hospital, the standard therapy given to post-craniotomy patients with mechanical ventilation is analgesic and sedation. This standard therapy is also given according to the patient's clinical condition

SUMMARY:
The aim of this clinical trial is to prove that acupuncture therapy combined with standard therapy can optimize hemodynamics and reduce pain in post-craniotomy patients with mechanical ventilation. The main questions it aims to answer are:

* Is there a difference in mean arterial pressure, pulse rate, respiratory rate, oxygen fraction and pain in the acupuncture therapy group combined with standard therapy compared to standard therapy after the 3rd therapy and compared to before therapy?
* Is there a difference in changes in ventilator mode in the acupuncture therapy group combined with standard therapy compared to standard therapy after the 3rd therapy?
* Are there any side effects in the acupuncture therapy group combined with standard therapy?

Researchers will compare acupuncture therapy combined with standard therapy to standard therapy only

Participants will:

* receive acupuncture therapy for 3 consecutive days
* outcomes will be assessed after 3 days of therapy.

DETAILED DESCRIPTION:
* Standard therapy is pharmacological therapy administered by the patient's attending anesthesiologist to research subjects in accordance with existing clinical practice guidelines. At the ICU of Tangerang District General Hospital, standard therapy administered to patients post-craniotomy with mechanical ventilation includes symptomatic therapy based on the patient's symptoms and condition (including antihypertensive medications, typically calcium channel blockers administered intravenously or orally), analgesics (typically fentanyl or morphine), and sedation (midazolam or propofol). This standard therapy is also administered according to the patient's clinical condition.
* Hemodynamic refers to parameters assess whether perfusion in the body is adequate or not, including how the heart pumps blood, how blood vessels carry blood throughout the body, and how blood nourishes and supplies oxygen to body tissues. Hemodynamic outcomes are assessed through vital signs such as blood pressure or Mean Arterial Pressure, pulse rate, respiratory rate, and oxygen requirements (FiO2).
* Critical Care Pain Observation Tools (CPOT) is a pain assessment tool for patients who are unable to communicate verbally and are on a ventilator. The assessment includes facial expressions, body movements, muscle tension, and compliance with the ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Subjects who received craniotomy with vascular etiology
* Conscious patients with GCS over 9 before craniotomy
* Using SIMV mode mechanical ventilation
* Family willing for the patient to participate in the study until completion and signed informed consent

Exclusion Criteria:

* History of neuromusculoskeletal diseases such as myasthenia gravis or multiple sclerosis
* Treatment for lung cancer and COVID-19
* There is infection, scarring or malignancy in the acupuncture stabbing area
* Patients with blood clotting disorders, platelets under 50. 000/µl, patients on anticoagulant therapy with INR over 2.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Pressure | Before therapy, Day 4
  Average arterial pressure during one cardiac cycle of systole and diastole
Heart Rate | Before therapy, Day 4
  Measurement of the participant's pulse rate over one minute.
Respiration Rate | Before therapy, Day 4
  Measurement of the participant's respiratory rate over one minute.
Oxygen Fraction | Before therapy, Day 4
  Oxygen concentration in the inhaled gas mixture, as displayed on the patient monitor.
Critical care Pain Observation Tools | Before therapy, Day 4
  Pain assessment in non-verbal and mechanically ventilated patients, including facial expressions, body movements, muscle tension, and compliance.

SECONDARY OUTCOMES:
Ventilator Mode | Day 4
  Changes in the type of ventilator settings used for the participant.
Side Effect | Day 4
  Patient-reported complaints after receiving manual acupuncture therapy.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — the Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No